CLINICAL TRIAL: NCT06333171
Title: 4-aminopyridine for Skin Wound Healing
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Elfar (Other)
Responsible Party: Sponsor-Investigator, John Elfar, Tenured Professor, Chairman, Department of Orthopaedic Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00003872
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Wounds; Wound of Skin; Wound Heal; Wounds and Injuries
Keywords: 4 aminopyridine; wound healing
MeSH Terms: conditions — Wounds and Injuries | interventions — 4-Aminopyridine

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled trial design.
Who Masked: Participant, Investigator
Masking Description: Subjects in both aims will be assigned to Group A or Group B using a randomization scheme. Each study participant for each aim is randomly assigned to either treatment of placebo using permuted block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: 4-aminopyridine (Active Comparator): dalfampridine (generic) 10 mg capsule po every 12 hours
  Interventions: Drug: 4-Aminopyridine
- Group B: Placebo (Placebo Comparator): Placebo-1 capsule po every 12 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 4-Aminopyridine — Active study drug
  Other Names: 4AP, dalfampridine
  Arms: Group A: 4-aminopyridine
Other: Placebo — Placebo comparator
  Arms: Group B: Placebo

SUMMARY:
Many patients suffer from chronic non-healing wounds as well as acute wounds. There is a need to develop treatments to accelerate and improve healing of chronic and acute wounds. More research is needed to evaluate the role of 4-aminopyridine (4-AP), a promising new agent with an excellent safety profile, on wound healing. The investigational treatment will be used to evaluate the role of (4-AP) on the treatment of wounds to accelerate wound healing in healthy adults.

The purpose of this study is to evaluate the role of 4-AP on the treatment of wounds to accelerate healing.

The investigational treatment will be used to test the hypothesis that 4-AP can speed wound healing.

DETAILED DESCRIPTION:
Worldwide, hundreds of millions of patients suffer from chronic non-healing wounds. In addition, most people will experience acute wounding at some point in their life. There is a need to develop agents to treat chronic and acute wounds. This need has intensified with the aging of the population, the rising incidence of diabetes and obesity, and the increasing number of patients undergoing treatment with medications that adversely affect wound healing.

Through experiments performed on animals with 4-aminopyridine, (currently marketed by Acorda Healthcare, Inc. in slow-release form as AMPYRA®, and available in generic form proposed for use in this study), the investigators found striking effects on wounds in the standard rodent model used in the literature. In these experiments, animals with wounds held open with stents, healed faster with mass-adjusted human doses of 4-AP. All relevant markers of tissue regeneration were augmented with 4-AP treatment. These injuries are considered standard models, used for decades that correlate to those encountered in the human patients.

The investigators found that:

1. 4-AP administration over just 21 days led to a large augmentation of wound healing at time points as early as three days post injury.
2. 4-AP treatment was associated with no adverse events in animals at the doses used consistent with our previous applications.
3. Numerous measures of wound healing at the cellular level showed quantifiable improvement with treatment at the tissue level.

4-AP is used in some of the most fragile of neurologically-ailing patients and is currently a mainline treatment in the setting of multiple sclerosis. Multiple sclerosis patients suffer a demyelinating disorder that causes the stripping of the myelin sheath from around neurons in the peripheral and central nervous system. The myelin covering allows for normal conduction of impulses and, without such covering, impulses are small, impaired, impeded, and ineffective. The recognition that crush injuries to nerves do not simply sever the axonal fibers but also demyelinate some population of nerve cells has led to the idea to study the treatment of peripheral nerve traumatic injuries in humans using 4-AP and this continues to be the subject of some of the investigator's other translational work

There is extant literature demonstrating the positive effects of electrical stimulation in wound healing. Electrical stimulation of wounds has been shown to be effective in accelerating wound repair for diabetic foot ulcers and other chronic skin ulcers. Direct electrical stimulation of the skin is labor intensive, while 4-AP is more easily administered as an oral therapy. Thus, the recognition that re-innervation may improve healing in the wound bed - and that 4-AP has a differential, clinically relevant effect on nerves and wounds naturally leads to this application.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy adult patients without skin conditions effecting the skin of the axilla or upper inner arm.
* Cognitive ability to evaluate wound healing, report sensory and motor deficit during examination.
* Eligible for standard of care plan for wound closure by secondary intention (normal healing without intervention).
* Adults subject aged 18-70
* Ability to give written informed consent.
* Capable of safely coming in for follow up visits on all scheduled appointments.

Exclusion Criteria:

* History of multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of hypersensitivity to AMPYRA® or 4-aminopyridine
* Current use of aminopyridine medications, including other compounded 4-AP
* Suspected renal impairment based on the Choyke questionnaire.
* History of difficult compliance with timely follow up
* Patients outside the age range
* Unable to provide informed consent.
* Patients with a known history of a seizure disorder (4-AP overdose can, in selected cases, result in limited seizure activity).
* Patients with a concomitant traumatic brain injury.
* Patients unable to communicate.
* Patients unwilling to complete the study requirements.
* Patients currently taking organic cat-ion transporter 2 (OCT2) inhibitors, e.g. Cimetidine.
* Pregnancy, breastfeeding or incarcerated individuals.
* Non-English speaking
* Patients unable or unwilling to take calibrated (with gauge) photographs of their wounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Return of skin integrity and wound closure after skin punch biopsy | 6 weeks
  Axillary skin punch biopsies will be performed on healthy volunteers. Wound healing will be measured using visual assessment.

SECONDARY OUTCOMES:
The effect of 4-AP on the hair number and growth at the skin punch biopsy site. | 6 weeks
  The axillary skin punch biopsies will evaluated for the number of hair follicles and hair growth.

CONTACTS AND LOCATIONS:
Overall Officials: John Elfar, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.